CLINICAL TRIAL: NCT01625026
Title: Effects of Obeticholic Acid on Hepatic Fatty Acid/Triglyceride Metabolism and Hepatobiliary Detoxification/Elimination in Morbidly Obese and Gallstone Patients
Brief Title: Obeticholic Acid in Bariatric and Gallstone Disease
Acronym: OCABSGS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Hanns-Ulrich Marschall, Professor of Clinical Hepatology, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OCABSGS
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Obesity; Gallstones
Keywords: Morbidly obesity; Gastric bypass; Cholecystolithiasis
MeSH Terms: conditions — Obesity; Gallstones; Cholecystolithiasis | interventions — obeticholic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Morbid Obesity OCA (Active Comparator): Obeticholic acid 25 mg/day in three weeks
  Interventions: Drug: Obeticholic acid
- Morbid Obesity Placebo (Placebo Comparator): Obeticholic acid 25 mg/day matching placebo in three weeks
  Interventions: Drug: Placebo
- Gallstones OCA (Active Comparator): Obeticholic acid 25 mg/day in three weeks
  Interventions: Drug: Obeticholic acid
- Gallstones Placebo (Placebo Comparator): Obeticholic acid 25 mg/day matching placebo in three weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Obeticholic acid — Obeticholic acid 25 mg/day in three weeks
  Other Names: INT-747
  Arms: Gallstones OCA; Morbid Obesity OCA
Drug: Placebo — Placebo to obeticholic acid
  Other Names: Placebo INT-747
  Arms: Gallstones Placebo; Morbid Obesity Placebo

SUMMARY:
By binding to the nuclear receptor FXR, bile acids not only regulate their own turn-over but presumably also pivotal steps in cholesterol, triglyceride and glucose metabolism as shown in laboratory animals. Obeticholic acid (OCA) is a semisynthetic bile acid with very high affinity to FXR. In a pharmacodynamic study the effects of OCA on bile acid, lipid and glucose turn-over are studied in 20 morbidly obese and 20 gallstones patents, respectively, that are administered OCA at 25 mg/day in three weeks before bariatric (BS) or gallstone (GS) surgery where in addition to blood samples also biopsies are taken from the liver and in the case of BS, omental and subcutaneous adipose tissue and in case of GS, gallbladder bile.

DETAILED DESCRIPTION:
In a placebo-controlled double-blind randomized trial, 20 otherwise healthy morbidly obese patients scheduled for bariatric surgery, and 20 otherwise healthy gallstone patients will be administered 25 mg/day INT-747 or placebo for three weeks until the day before surgery. Serum from days 1 and 21 will be analyzed for routine liver tests, bile acids, a complete lipid profile including FA and in addition for 7α-hydroxy-4-cholesten-3-one and FGF-19, markers for bile acid synthesis and its intestinal stimulation. For the evaluation of insulin resistance and possible pre-diabetes, plasma will be taken for the estimation of HOMA index and oral glucose tolerance test (OGTT) will be performed at days 1 and 21. At surgery, a liver biopsy (0.5-1 g) and a white adipose tissue (WAT) specimen (1 cm2) will be taken and immediately frozen in liquid nitrogen for mRNA and protein preparation for quantitative RT-PCR and Western analysis, respectively, histopathological NAFLD grading, and measuring of hepatic and WAT lipase activity. In gallstone patients, gallbladder bile will be sampled for the measurements of biliary lipids (cholesterol, phospholipids, bile acids) and the calculation of the cholesterol saturation index.

ELIGIBILITY:
Inclusion Criteria:

* In the obesity group: BMI ≥35 kg/m2
* In the gallstone group: symptomatic, ultrasound verified gallstone disease

Exclusion Criteria:

* Chronic liver disease other than NAFLD (viral hepatitis, autoimmune liver disease, hemochromatosis, homozygous alpha1-antitrypsin deficiency and Wilson disease)
* Previous gastric or small bowel surgery
* Inflammatory bowel disease
* Uncontrolled diabetes mellitus (fasting blood glucose >6.7 mmol/L), hypothyroidism or hyperthyroidism, or other significant endocrine disease.
* Pregnancy. A urine pregnancy test will be performed the day before start of medication. Women of childbearing potential can only be included if a safe and reliable contraception is used, e.g., oral contraceptives.
* Elevations of transaminases (ALAT/ASAT) or alkaline phosphatase or bilirubin above 2xULN (upper limit of normal) the day before start of medication.
* Other serious disease, including depressive disorders treated by medication
* Patients who will not comply with the protocol.
* A subject who is euthyroid on a stable replacement dose of thyroid hormone is acceptable provided the TSH is within normal range.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Effects of OCA on FXR-dependent metabolism | Day 21
  Primary endpoints
  * relative changes in markers for insulin resistance
  * relative changes in FA and TG
  * relative changes in hepatic and adipose tissue lipase expression and activity
  * relative changes in hepatic apical transport proteins ABCG5/8, BSEP, MDR3, MRP2
  * relative changes in hepatic ER stress markers

SECONDARY OUTCOMES:
Effects of OCA on serum lipid levels | 21 days
  Secondary endpoints
  * relative changes in m RNA expression levels of genes listed under 3.ix
  * relative changes in hepatic basolateral transport proteins listed under 3.x
  * relative change in serum bile acids as listed under 3.xii, including INT-747
  * relative changes in biliary lipids (cholesterol, phospholipids, bile acids)
  * relative change in plasma 7α-hydroxy-4-cholesten-3-one and FGF-19
  * relative changes in total cholesterol, LDL-C, HDL-C, Apo A1, Apo B, in Lp(A)

CONTACTS AND LOCATIONS:
Overall Officials: Hanns-Ulrich Marschall, MD, PhD, Principal Investigator — Sahlgrenska University Hospital Gothenburg
Locations (1):
- Hanns-Ulrich Marschall, Gothenburg, Sweden

REFERENCES:
- [Derived] Al-Dury S, Wahlstrom A, Panzitt K, Thorell A, Stahlman M, Trauner M, Fickert P, Backhed F, Fandriks L, Wagner M, Marschall HU. Obeticholic acid may increase the risk of gallstone formation in susceptible patients. J Hepatol. 2019 Nov;71(5):986-991. doi: 10.1016/j.jhep.2019.06.011. Epub 2019 Jun 27. PMID 31254596